CLINICAL TRIAL: NCT00821496
Title: A Phase I, Open Label, Fixed Sequence, Single-Center Study to Evaluate the Effect of Multiple Dose Administration of VI-0521 on the Pharmacokinetics of a Single Dose of Oral Contraceptive in Healthy Female Subjects
Brief Title: Evaluate the Effect of VI-0521 on the Pharmacokinetics of Oral Contraceptive in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB-108
Record Dates: First submitted 2009-01-06; First posted 2009-01-13 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Multiple dose administration; Oral Contraceptives
MeSH Terms: interventions — Ethinyl Estradiol; Norethindrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Contraceptive (Experimental)
  Interventions: Drug: ethinyl estradiol, norethindrone, VI-0521

INTERVENTIONS:
Drug: ethinyl estradiol, norethindrone, VI-0521 — Oral contraceptive
  Other Names: VI-0521, Ortho-Novum 1/35-28

SUMMARY:
This study is desgigned to look at the effect of multiple dosing administration of VI-0521 on Oral Contraceptive medication.

DETAILED DESCRIPTION:
This study is designed to determine if multiple oral doses of VI-0521 would alter the pharmacokinetics of an oral contraceptive in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Females, 19 - 64 years of age (inclusive), who are non-pregnant, not planning pregnancy and non-breast-feeding.
2. If females of child-bearing potential, be using adequate contraception, defined as double barrier methods, single barrier plus tubal ligation.
3. A body weight of at least 50 kg and a body mass index (BMI) between 27 and 35 kg/m2, inclusive.
4. Medically healthy, with clinically insignificant screening results.
5. Subjects are able to communicate with the investigator, and to understand and comply with all requirements of study participation.
6. Voluntarily consent to participate in the study.

Exclusion Criteria:

1. A history or presence of significant cardiovascular, neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the investigator.
2. Any clinically significant laboratory abnormalities as judged by the investigator.
3. Any history of glaucoma, increased intraocular pressure, or medications to treat increased intraocular pressure.
4. Presence of cholelithiasis or cholecystitis within the last 6 months that has not been surgically treated with cholecystectomy.
5. Any history of a cardiovascular or cerebrovascular event.
6. Systolic blood pressure > 150 mm Hg or diastolic blood pressure > 95 mm Hg at screening or at check-in on Day -1.
7. Positive urine drug test, serum cotinine test, pregnancy test and/or positive urine alcohol test at screening or check in Day -1.
8. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening.
9. Any history or presence of alcoholism or drug or substance abuse as defined by the investigator.
10. Any active malignancy except basal cell carcinoma.
11. A history of breast cancer.
12. Any history of bipolar disorder or psychosis, history of psychiatric hospitalization, greater than one lifetime episode of major depression.
13. A history of intolerance to oral contraceptives.
14. A history of hypersensitivity or idiosyncratic reaction to the active drugs, compounds related to the study drugs or to any excipients present in the VI-0521 capsule.
15. Use of any prescription or over-the-counter (OTC) medication, including herbal products, within the 14 days prior to Day -1. Up to 2 g per day of acetaminophen is allowed at the discretion of the Investigator.
16. Use of any drug known to have a significance in inhibiting or inducing liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to Day -1.
17. Blood donation or significant blood loss within 56 days prior to Day -1.
18. Plasma donation within 7 days prior to Day -1.
19. Any use of tobacco or nicotine products within 3 months prior to Day -1.
20. Any history of celiac diseases, food allergies, and those on vegetarian or other diets incompatible with study objectives.
21. Any subject who received an investigational drug within 30 days or six half-lives, whichever is longer, prior to dosing in this study.
22. Clinical judgment by the investigator that the subject should not participate in the study.
23. Involvement in the planning and conduct of the study.
24. Any subject who has participated in a previous clinical trial with VI-0521.
25. Subjects with any condition possibly affecting drug absorption.

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
PK of the Oral contraceptive agent | 31 days

SECONDARY OUTCOMES:
saftey and tolerability of multiple dose adminstration of VI-0521 in healthy female subjects | 31

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, Study Director — VIVUS LLC; Scott Sharples, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States